CLINICAL TRIAL: NCT07056322
Title: Optimal Meals to Reduce Bone Resorption in Women With Osteopenia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OsteoMeal-study1; PhD030-24 (Other Grant/Funding Number: Danish Diabetic and Endocrine Academy)
Record Dates: First submitted 2025-06-27; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Osteopenia
Keywords: Osteopenia; Meal intervention; Bone turnover
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Milk

STUDY DESIGN:
Intervention Model Description: The cross-over trial study consists of six study days, where the women in random order at 08.00 are administered a) 100 ml yoghurt natural b) 200 ml yoghurt natural, c) 100 ml of milk, d) 100 g banana e) dairy and fibers, and f) fasting. The participants will meet at 07.00 on the study days after an overnight fast. 24 hours before the study days the participants are asked to refrain from exercise and alcohol.
  During the study days blood samples are collected from an intravenous access hourly from 08.00 until 14.00 to measure changes in bone turnover markers and gut hormones.
Masking Description: Blinding of participants is not possible, laboratory staff who will analyse the blood samples, will be blinded to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meals or fasting in randomized order (Experimental): All participants will receive each of the six interventions (five different meals and one fasting control) in randomized order, with a minimum 1 week washout between test days. The order of the interventions is individually randomized. Blood samples will be collected at arrival and hourly during each visit to assess bone turnover markers.
  Interventions: Dietary Supplement: 200 ml dairy; Dietary Supplement: 100 ml milk; Dietary Supplement: 100 g banana; Dietary Supplement: 100 ml dairy and fibers; Other: Fasting (control); Dietary Supplement: 100 ml dairy

INTERVENTIONS:
Dietary Supplement: 200 ml dairy — Participants consume the meal after a fasting baseline bloodsample. Bloodsamples are collected over a six-hour period to evaluate postpandrial changes in bone turnover markers.
Dietary Supplement: 100 ml milk — Participants consume the meal after a fasting baseline bloodsample. Bloodsamples are collected over a six-hour period to evaluate postpandrial changes in bone turnover markers.
Dietary Supplement: 100 g banana — Participants consume the meal after a fasting baseline bloodsample. Bloodsamples are collected over a six-hour period to evaluate postpandrial changes in bone turnover markers.
Dietary Supplement: 100 ml dairy and fibers — Participants consume the meal after a fasting baseline bloodsample. Bloodsamples are collected over a six-hour period to evaluate postpandrial changes in bone turnover markers.
Other: Fasting (control) — Participants consume the meal after a fasting baseline bloodsample. Bloodsamples are collected over a six-hour period to evaluate postpandrial changes in bone turnover markers.
Dietary Supplement: 100 ml dairy — Participants consume the meal after a fasting baseline bloodsample. Bloodsamples are collected over a six-hour period to evaluate postpandrial changes in bone turnover markers.

SUMMARY:
The goal of this clinical trial is to investigate whether different types of small meals can help reduce bone loss in postmenopausal women with osteopenia, a condition where bone density is lower than normal and may lead to osteoporosis.

The main hypothesis is:

- A small amount of dairy (100 ml) is just as effective as a larger meal containing dairy and banana in reducing bone resorption.

Based on this, the study aims to answer the following questions:

- Which type and size of meal is most effective in reducing bone resorption?

Researchers will compare five different types of meals to a fasting control day to determine which meals best reduce markers of bone loss in the blood.

Participants will attend six clinical visits: five involving the intake of different test meals, and one control visit involving fasting. The participants will have blood samples taken over a period of 6 hours after each meal or fasting period to measure markers of bone metabolism.

This study aims to identify a simple, non-drug-based strategy to support bone health and help prevent progression to osteoporosis.

DETAILED DESCRIPTION:
This project investigates whether administration of a meal can reduce bone resorption and thereby, if used strategic, prevent the development of osteoporosis in postmenopausal women with osteopenia, as measured by bone turnover markers and bone density. Furthermore, it is investigated which type and size of meal is optimal for bone health in osteopenia.

The project comprises of one hypotheses:

- 100 ml dairy is as effective as larger amounts of dairy and banana in decreasing bone resorption.

Osteopenia is a prevalent condition and is a precursor to osteoporosis and fractures. In 2011 it is estimated that osteoporotic fractures resulted a total cost of 1.6 billion EUR in Denmark. Osteopenia is diagnosed by a low bone mineral density (BMD), with a T-score between -1.1 and - 2.4, whereas osteoporosis is diagnosed by a T-score of ≤2.5. In postmenopausal women, it is estimated that 43 % have osteopenia. The current recommendation to prevent fractures in osteopenia is sufficient intake of vitamin D and calcium, besides smoking cessation, physical activity, and moderate alcohol intake. In case of osteoporosis, additional anti-osteoporotic medications are recommended, which have been shown to reduce fracture rates. However, effective non-pharmacologic remedies to prevent progression from osteopenia to osteoporosis are urgently needed and the potential of timing of meals in this context should therefore be explored. Osteopenia and osteoporosis are caused by an increased bone resorption to bone formation ratio which decreases BMD and increases fractures. During the bone resorption and bone formation phases; products are released to the bloodstream and can be measured as bone turnover markers. Carboxy-terminal collagen crosslinks (CTX) is a bone resorption marker and procollagen type I Npropeptide (P1NP) is a bone formation marker and they are internationally recommended as the standard bone turnover markers. Following a meal, bone resorption decreases. The gut hormone; glucagon-like peptide 2 (GLP-2) is released to the circulation following a meal and reduces bone resorption, as measured by CTX, by 50 %. In humans bone resorption is highly increased during the night time (fasting state) and gut hormones have therefore been suggested as treatments for osteoporosis. In a previous study, GLP-2 was administered subcutaneously before bedtime for 120 days and showed a decrease in nightly CTX levels and an increase in bone mineral density at the hip and no signs of tachyphylaxis during the treatment. The investigators have shown that a meal suppresses CTX levels for as long as six hours with a simultaneous increase in GLP-2 and that the oral administration of nutrients is essential for a reduction in CTX. The investigators have great experience in conducting clinical trials assessing bone health. In this project it is investigated which type and size of meals reduce CTX most profoundly.

The meals in this study are selected as 3.5 % fatty dairy or banana as these are commonly used smaller meals. Furthermore, the gastric emptying of a dairy depends on the meal size, and fat reduces the gastric emptying, whereas banana contains fibers and may thus have a shorter gastric emptying. Yoghurt is expected to have slower gastric emptying than milk primarily due to its higher viscosity. Additionally yoghurt is a more fermented product compared to milk, potentially affecting the postprandial gut hormone response differently. Psyllium and banana (pectin fibers) are both dietary fiber sources but differ in fiber composition and solubility, which may lead to different effects on gastric emptying and gut hormone responses. The fiber content differs between banana and psyllium, with psyllium being more concentrated. We aim to adjust the fiber content to be approximately equivalent, so participants will receive 4-5 g of psyllium (1 teaspoon), providing about the same amount of fiber as 100 g of banana.

The results from this study will be used for a follow up study in which the effects on bone health of meal administration over a longer period will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Osteopenia at the lumbar spine defined as BMD t-score -2.4 to -1.1.
* Postmenopausal women
* Age < 80 years
* CTX level ≥ 0.40 ng/ml
* BMI 17-25 kg/m2

Exclusion Criteria:

* A diagnosis of osteoporosis, diabetes, primary hyperparathyroidism or active malignancy.
* Current or recent (within two years) use of systemic glucocorticoids for 4 continuous weeks or more, anticonvulsants or anti-osteoporotic drugs including systemic estrogen treatment.
* Low p-25-OH vitamin D-levels (< 50 pmol/l)
* Estimated glomerular filtration (eGFR) <60 ml/min

Max Age: 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Bone resoroption | From enrollment through six study visits over a period of approximately 12 weeks
  The primary endpoint of the study is difference in the area under curve of the bone resorption marker CTX during the different study days

SECONDARY OUTCOMES:
Change in bone formation marker P1NP | From enrollment through six study visits over a period of approximately 12 weeks
  Secondary outcome assesing changes in the bone formation marker P1NP
Changes in osteocalcin levels | From enrollment through six study visits over a period of approximately 12 weeks
  Secondary outcome assesing changes in the bone turnover marker osteocalcin
Changes in immune respons (Treg/Th17 cell ratio) | From enrollment through six study visits over a period of approximately 12 weeks
  Secondary outcome assesing changes in the immune cell composition (Treg/Th17 cell ratio)
Changes in the incretin hormone GLP-2 | From enrollment through six study visits over a period of approximately 12 weeks
  Secondary outcome assesing changes in levels of GLP-2

CONTACTS AND LOCATIONS:
Overall Officials: Jakob S Linde, Medical Doctor, MD, PhD, Principal Investigator — Department of Endocrinology and Internal Medicine, Aarhus University Hospital
Locations (1):
- Department of Endocrinology and Internal Medicine, Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Giuntini EB, Sarda FAH, de Menezes EW. The Effects of Soluble Dietary Fibers on Glycemic Response: An Overview and Futures Perspectives. Foods. 2022 Dec 6;11(23):3934. doi: 10.3390/foods11233934. PMID 36496742
- [Background] Weber AM, Pascale N, Gu F, Ryan EP, Respondek F. Nutrition and health effects of pectin: A systematic scoping review of human intervention studies. Nutr Res Rev. 2025 Jun;38(1):306-323. doi: 10.1017/S0954422424000180. Epub 2024 Sep 26. PMID 39324277
- [Background] Sanggaard KM, Holst JJ, Rehfeld JF, Sandstrom B, Raben A, Tholstrup T. Different effects of whole milk and a fermented milk with the same fat and lactose content on gastric emptying and postprandial lipaemia, but not on glycaemic response and appetite. Br J Nutr. 2004 Sep;92(3):447-59. doi: 10.1079/bjn20041219. PMID 15469648
- [Background] Ring J, Sharkoff D, Richter W. Intravascular persistence of hydroxyethyl starch (HES) after serial granulocyte collections using HES in man. Vox Sang. 1980 Oct;39(4):181-5. doi: 10.1111/j.1423-0410.1980.tb01855.x. PMID 6163255
- [Background] Berry SD, McLean RR, Hannan MT, Cupples LA, Kiel DP. Changes in bone mineral density may predict the risk of fracture differently in older adults according to fall history. J Am Geriatr Soc. 2014 Dec;62(12):2345-9. doi: 10.1111/jgs.13127. Epub 2014 Nov 29. PMID 25438807
- [Background] Sayon-Orea C, Martinez-Gonzalez MA, Ruiz-Canela M, Bes-Rastrollo M. Associations between Yogurt Consumption and Weight Gain and Risk of Obesity and Metabolic Syndrome: A Systematic Review. Adv Nutr. 2017 Jan 17;8(1):146S-154S. doi: 10.3945/an.115.011536. Print 2017 Jan. PMID 28096138
- [Background] Miller KC. Plasma potassium concentration and content changes after banana ingestion in exercised men. J Athl Train. 2012 Nov-Dec;47(6):648-54. doi: 10.4085/1062-6050-47.6.05. PMID 23182013
- [Background] Keszthelyi D, Knol D, Troost FJ, van Avesaat M, Foltz M, Masclee AA. Time of ingestion relative to meal intake determines gastrointestinal responses to a plant sterol-containing yoghurt drink. Eur J Nutr. 2013 Jun;52(4):1417-20. doi: 10.1007/s00394-012-0440-3. Epub 2012 Aug 23. PMID 22915051
- [Background] Starup-Linde J, Ornstrup MJ, Kjaer TN, Lykkeboe S, Handberg A, Gregersen S, Harslof T, Pedersen SB, Vestergaard P, Langdahl BL. Bone Density and Structure in Overweight Men With and Without Diabetes. Front Endocrinol (Lausanne). 2022 Mar 10;13:837084. doi: 10.3389/fendo.2022.837084. eCollection 2022. PMID 35360074
- [Background] Fuglsang-Nielsen R, Rakvaag E, Vestergaard P, Hermansen K, Gregersen S, Starup-Linde J. The Effects of 12-Weeks Whey Protein Supplements on Markers of Bone Turnover in Adults With Abdominal Obesity - A Post Hoc Analysis. Front Endocrinol (Lausanne). 2022 Mar 29;13:832897. doi: 10.3389/fendo.2022.832897. eCollection 2022. PMID 35422766
- [Background] Veldhuis-Vlug AG, Rosen CJ. Mechanisms of marrow adiposity and its implications for skeletal health. Metabolism. 2017 Feb;67:106-114. doi: 10.1016/j.metabol.2016.11.013. Epub 2016 Nov 27. PMID 28081773
- [Background] Westberg-Rasmussen S, Starup-Linde J, Hermansen K, Holst JJ, Hartmann B, Vestergaard P, Gregersen S. Differential impact of glucose administered intravenously or orally on bone turnover markers in healthy male subjects. Bone. 2017 Apr;97:261-266. doi: 10.1016/j.bone.2017.01.027. Epub 2017 Jan 23. PMID 28126633
- [Background] Henriksen DB, Alexandersen P, Hartmann B, Adrian CL, Byrjalsen I, Bone HG, Holst JJ, Christiansen C. Four-month treatment with GLP-2 significantly increases hip BMD: a randomized, placebo-controlled, dose-ranging study in postmenopausal women with low BMD. Bone. 2009 Nov;45(5):833-42. doi: 10.1016/j.bone.2009.07.008. Epub 2009 Jul 22. PMID 19631303
- [Background] Bjarnason NH, Henriksen EE, Alexandersen P, Christgau S, Henriksen DB, Christiansen C. Mechanism of circadian variation in bone resorption. Bone. 2002 Jan;30(1):307-13. doi: 10.1016/s8756-3282(01)00662-7. PMID 11792602
- [Background] Bjornshave A, Lykkeboe S, Hartmann B, Holst JJ, Hermansen K, Starup-Linde J. Effects of a whey protein pre-meal on bone turnover in participants with and without type 2 diabetes-A post hoc analysis of a randomised, controlled, crossover trial. Diabet Med. 2021 Jun;38(6):e14471. doi: 10.1111/dme.14471. Epub 2020 Dec 13. PMID 33259643
- [Background] Vasikaran S, Cooper C, Eastell R, Griesmacher A, Morris HA, Trenti T, Kanis JA. International Osteoporosis Foundation and International Federation of Clinical Chemistry and Laboratory Medicine position on bone marker standards in osteoporosis. Clin Chem Lab Med. 2011 Aug;49(8):1271-1274. doi: 10.1515/CCLM.2011.602. Epub 2011 May 24. PMID 21605012
- [Background] Shoback D, Rosen CJ, Black DM, Cheung AM, Murad MH, Eastell R. Pharmacological Management of Osteoporosis in Postmenopausal Women: An Endocrine Society Guideline Update. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgaa048. doi: 10.1210/clinem/dgaa048. PMID 32068863
- [Background] Hansen L, Mathiesen AS, Vestergaard P, Ehlers LH, Petersen KD. A health economic analysis of osteoporotic fractures: who carries the burden? Arch Osteoporos. 2013;8(1):126. doi: 10.1007/s11657-013-0126-3. Epub 2013 Feb 19. PMID 23420317
- [Background] Guzman Ibarra M, Ablanedo Aguirre J, Armijo Delgadillo R, Garcia Ruiz Esparza M. [Prevalence of osteopenia and osteoporosis assessed by densitometry in postmenopausal women]. Ginecol Obstet Mex. 2003 May;71:225-32. Spanish. PMID 12908337